CLINICAL TRIAL: NCT05322083
Title: Analysis of HIV Subtype A6 Genome in Patients With Virological Failure After Switching to Doravirine (DOR)
Brief Title: HIV A6 Genome In ART Unsuccessful Patients On DOR
Acronym: HIV-A6-DOR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: MSD Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MISP#60102
Record Dates: First submitted 2022-03-22; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Virus-HIV
Keywords: HIV, mutation, resistance
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — doravirine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma and whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- HIV patients: All patients will be prescribed treatment drugs in accordance with the national protocol by the doctors of the AIDS centers. The decision to prescribe Doravirine will also be made by doctors.
  Interventions: Drug: Doravirine

INTERVENTIONS:
Drug: Doravirine — Doravirine will be given to patients after failure on the first NNRTI regimen.
  Other Names: DOR

SUMMARY:
The aim of the study is to evaluate the efficacy of Doravirine (DOR) in the second-line therapy for patients infected with HIV-1 sub-subtype A6 and its derivatives and having the mutations to previously used drugs

DETAILED DESCRIPTION:
During the study 60-80 HIV-infected patients in 2-4 investigation sites (AIDS Centers) across Russia with proven virological failure on first-line antiretroviral therapy (ART) including efavirenz (EFV) and nevirapine (NVP) will be enrolled. The blood samples, epidemiological, clinical and demographic data of patients participating in the study must be collected. All participants must provide written informed consent before the start of the study.

Virological failure on NNRTI regimen in all the participants will be confirmed by HIV genotyping. All the patients with confirmed NNRTI mutations will be switched to DOR instead of EFV/NVP in the second-line therapy and enrolled to the study.

The primary efficacy endpoints of ART with DOR will be weeks 8 and 24 (viral load + T-cell count). For all samples with virological failure at weeks 8 or 24 HIV-1 DNA sequences (full protease (PR) and partial reverse transcriptase (RT) regions) will be obtained using the in-house test system or commercial kit (Central Research Institute of Epidemiology, Moscow, Russia). In case of virological failure of DOR treatment, the analysis of drug resistance mutations will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection confirmed
* > 18 years
* Informed consent signed

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult (over 18 years of age) patients who have a confirmed diagnosis of HIV infection will be invited to participate in the study. Military personnel and pregnant women will not be included in the study unless such studies are necessary for these patients. Patients must have a virologic failure on their first ART regimen that includes NNRTIs.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
HIV viral load | Week 8
  The result of measuring the HIV viral load 8 weeks after the start of DOR-based treatment. The success of therapy will correspond to an undetectable level of viral load (less than 50 RNA copies/ml) or a decrease of two logarithms compared with the values before treatment start. Upon receipt of a detected viral load, treatment will be nevertheless continued up to 24 weeks.
HIV viral load | Week 24
  The result of measuring the HIV viral load 24 weeks after the start of DOR-based treatment. The success of therapy will correspond to an undetectable level of viral load (less than 50 RNA copies/ml). Upon receipt of any detected viral load, the treatment will be considered a failure and the reasons for the failure (lack of adherence, drug interactions, non-compliance with dietary requirements, etc.) will be analyzed. If these causes are excluded, the HIV genotype will be analyzed for the presence of drug resistance mutations (RT genome region).

SECONDARY OUTCOMES:
HIV genotype | Week 24
  HIV genotype in patients experienced failure on DOR-based treatment regimen (RT genome region). The study of the genotype will make it possible to understand to which of the components of the therapy regimen the virus has developed resistance and which of the drugs needs to be replaced. If it turns out to be a drug from the basic regimen (not DOR but NRTIs), the regimen will be changed at the discretion of the attending physician (this decision is not within the scope of this project). If DOR resistance mutations are detected such as V106I or Y188L, their frequency will be estimated (the proportion of patients with such mutations ) and the spectrum of associated mutations will be analysed.

REFERENCES:
- [Background] Ayitewala A, Kyeyune F, Ainembabazi P, Nabulime E, Kato CD, Nankya I. Comparison of HIV drug resistance profiles across HIV-1 subtypes A and D for patients receiving a tenofovir-based and zidovudine-based first line regimens in Uganda. AIDS Res Ther. 2020 Jan 31;17(1):2. doi: 10.1186/s12981-020-0258-7. PMID 32005262
- [Background] Lapovok I, Laga V, Kazennova E, Bobkova M. HIV Type 1 Integrase Natural Polymorphisms in Viral Variants Circulating in FSU Countries. Curr HIV Res. 2017 Nov 23;15(5):318-326. doi: 10.2174/1570162X15666170815162052. PMID 28814231
- [Result] Baryshev PB, Bogachev VV, Gashnikova NM. Genetic characterization of an isolate of HIV type 1 AG recombinant form circulating in Siberia, Russia. Arch Virol. 2012 Dec;157(12):2335-41. doi: 10.1007/s00705-012-1442-4. Epub 2012 Aug 19. PMID 22903393
- [Result] Venner CM, Nankya I, Kyeyune F, Demers K, Kwok C, Chen PL, Rwambuya S, Munjoma M, Chipato T, Byamugisha J, Van Der Pol B, Mugyenyi P, Salata RA, Morrison CS, Arts EJ. Infecting HIV-1 Subtype Predicts Disease Progression in Women of Sub-Saharan Africa. EBioMedicine. 2016 Nov;13:305-314. doi: 10.1016/j.ebiom.2016.10.014. Epub 2016 Oct 12. PMID 27751765
- See also: Clinical Guidelines on treatment HIV-infection in Russia, 2017 — http://rushiv.ru/category/docs/national-recs/